CLINICAL TRIAL: NCT06157645
Title: Prophylactic Onlay Mesh Reinforcement vs Anatomical Closure in Stoma Reversal: A Randomized Controlled Trial
Brief Title: Prophylactic Mesh Reinforcement for Stoma Closure
Acronym: OASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelwahed Abdeljaber, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mesh with stoma closur
Record Dates: First submitted 2023-11-26; First posted 2023-12-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Incisional Hernia; Surgical Site Infection; Postoperative Pain; Hospital Stay, Length of Stay in Hospital From Surgery to Discharge; Complication
Keywords: Stoma closure; Stoma reversal; Loop ileostomy; Prophylactic mesh; Onlay mesh; Incisional hernia; Abdominal wall reinforcement; Anatomical closure; Randomized controlled trial; Surgical outcomes
MeSH Terms: conditions — Incisional Hernia; Surgical Wound Infection; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two parallel groups. The intervention group undergoes stoma reversal with prophylactic onlay Prolene mesh reinforcement, while the control group undergoes standard anatomical closure without mesh. Each participant receives only one assigned surgical technique, and outcomes are compared between the two groups.
Masking Description: This is an open-label study. Neither the participants, the treating surgeons, nor the outcome assessors are blinded to the assigned intervention due to the surgical nature of the procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): 1. Good preparation of the patient preoperative
  2. Performing an opening in the skin surrounding the stoma 3-4 mm from the muco-cutaneous junctions.
  3. Separate the bowel loop away from its attachment to the abdomen wall.
  4. Cut out a rim of 0.3-0.4 cm of scarred bowel edges exposes healthful tissue.
  5. Avoid any spillage or soiling
  6. Closing of bowel defect can be made by double layer of 3-0 vicryl interrupted.
  7. Once the tissue is of poor quality for simply closing, we expand the incision in the abdomen wall and resect a section. An end-to-end anastomosis is created using the conventional 2-layers suture method.
  8. Reduction of the bowel into the abdomen are carried out.
  9. irrigation the surgical field with a dilute anti-biotics or antiseptics and closure of the defect by continuous sutures using vicryl or prolene sutures
  10. Closure of the wound
- Group B (Experimental): 1. Good preparation of the patient preoperative
  2. Performing an opening in the skin surrounding the stoma 3-4 mm from the muco-cutaneous junctions.
  3. Separate the bowel loop away from its attachment to the abdomen wall.
  4. Cut out a rim of 0.3-0.4 cm of scarred bowel edges exposes healthful tissue.
  5. Avoid any spillage or soiling
  6. Closing of bowel defect can be made by double layer of 3-0 vicryl interrupted.
  7. Once the tissue is of poor quality for simply closing, we expand the incision in the abdomen wall and resect a section. An end-to-end anastomosis is created using the conventional 2-layers suture method.
  8. Reduction of the bowel into the abdomen are carried out.
  9. irrigation the surgical field with a dilute anti-biotics or antiseptics and closure of the defect by continuous sutures using vicryl or prolene sutures
  10. mesh is simply fixed over the defect as a tension-free patch (onlay)
  11. Closure of the wound
  Interventions: Device: Prolene mesh

INTERVENTIONS:
Device: Prolene mesh — Application of mesh onlay post stoma closure
  Arms: Group B

SUMMARY:
In the current work we are aiming to compare between the mesh-reinforced stoma closure and the anatomical closure in terms of the risk of developing surgical site incisional hernia (SSIH),incidence of surgical site infection , post-operative Pain and Hospital stay

DETAILED DESCRIPTION:
Intestinal stomas are used to divert intestinal content as a treatment option. Faecal flow is diverted from the site of the pathology by bringing the end or a loop of bowel through the anterior abdominal wall; any segments of the colon can be used, as well as the distal part of the ileum. A stoma may be temporary or permanent according to the condition. Temporary stomas are usually followed by elective stoma closure 6-8 weeks after. Though considered a relative safe procedure, studies reported high morbidity rates following stoma closure with different complications.

Incisional hernia following stoma closure occurs in up to 30% of patients. Incisional hernia affects quality of life, in regards to pain, physical function, ability to work, and cosmoses. Other serious complications due to bowel obstruction with incarceration or strangulation can occur which may necessitate reoperation. Mesh-reinforced stoma closure shown to decrease the incidence of surgical site incisional hernia (SSIH) with low complications risk. Though there is a debate about its efficacy due to lake of data ,and doubt to use a mesh in contaminated wounds due to fear of wounds complications which may necessitate mesh extraction or longer hospital stay make it hard for many surgeons to use Mesh-reinforced stoma closure.

In the current work we are aiming to compare between the mesh-reinforced stoma closure and the anatomical closure in terms of the risk of developing (SSIH),incidence of surgical site infection ,post-operative Pain and Hospital stay

ELIGIBILITY:
Inclusion Criteria:

* Patients who are fit for aesthesia.
* Patients with temporary double barrelled and simple loop ostomy
* Patients older than 16 years old

Exclusion criteria:

* Patients with end ostomy
* Infected stomas

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Incisional (stoma-site) hernia rate | Up to 12 months postoperatively
  Proportion of participants developing an incisional hernia at the stoma site, confirmed by physical examination or imaging (ultrasound/CT).

SECONDARY OUTCOMES:
Surgical site infection rate | Within 30 days postoperatively
  Rate of postoperative infections at the stoma closure site
post-operative Pain | Daily for the first 7 postoperative days
  Pain at the stoma closure site measured using the Visual Analog Scale (VAS).
Length of hospital stay | through study completion, an average of 2 years
  Number of days spent in hospital following surgery.
Postoperative complications | Within 30 days postoperatively
  Any postoperative complications, including wound dehiscence, ileus, bowel obstruction, or reoperation, graded according to Clavien-Dindo classification.
Operative time | Intraoperative (from skin incision to skin closure)
  Total duration of surgery measured in minutes.
Intraoperative blood loss | through study completion, an average of 2 years
  During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Thabet, Professor, Study Chair — Assiut University
Locations (1):
- Assiut university hospitals, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Background] Chow A, Tilney HS, Paraskeva P, Jeyarajah S, Zacharakis E, Purkayastha S. The morbidity surrounding reversal of defunctioning ileostomies: a systematic review of 48 studies including 6,107 cases. Int J Colorectal Dis. 2009 Jun;24(6):711-23. doi: 10.1007/s00384-009-0660-z. Epub 2009 Feb 17. PMID 19221766
- [Background] Williams NS, Nasmyth DG, Jones D, Smith AH. De-functioning stomas: a prospective controlled trial comparing loop ileostomy with loop transverse colostomy. Br J Surg. 1986 Jul;73(7):566-70. doi: 10.1002/bjs.1800730717. PMID 3524742
- [Background] Reinforcement of Closure of Stoma Site (ROCSS) Collaborative and the West Midlands Research Collaborative. Randomized controlled trial of standard closure of a stoma site vs biological mesh reinforcement: study protocol of the ROCSS trial. Colorectal Dis. 2018 Feb;20(2):O46-O54. doi: 10.1111/codi.13997. PMID 29314655
- [Background] Mohamedahmed AYY, Stonelake S, Zaman S, Hajibandeh S. Closure of stoma site with or without prophylactic mesh reinforcement: a systematic review and meta-analysis. Int J Colorectal Dis. 2020 Aug;35(8):1477-1488. doi: 10.1007/s00384-020-03681-0. Epub 2020 Jun 25. PMID 32588121
- [Background] Liu DS, Banham E, Yellapu S. Prophylactic mesh reinforcement reduces stomal site incisional hernia after ileostomy closure. World J Surg. 2013 Sep;37(9):2039-45. doi: 10.1007/s00268-013-2109-3. PMID 23716028
- [Background] Lee JH, Ahn BK, Lee KH. Complications Following the Use of Biologic Mesh in Ileostomy Closure: A Retrospective, Comparative Study. Wound Manag Prev. 2020 Jun;66(6):16-22. PMID 32511101